CLINICAL TRIAL: NCT06754969
Title: Does RPNI Reduce Incidence of Neuroma Formation Following Sural Nerve Biopsy: a Pilot Study
Brief Title: Does RPNI Reduce Incidence of Neuroma Formation Following Sural Nerve Biopsy
Acronym: NBxPilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Danielle Cohen, Resident, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H24-03129
Record Dates: First submitted 2024-10-22; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Neuroma of Lower Limb
Keywords: Sural Nerve Biopsy; Regenerative Peripheral Nerve Biopsy; RPNI
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be unaware whether they undergo sural nerve and muscle biopsy alone vs sural nerve, muscle biopsy, and RPNI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biopsy Alone (Active Comparator): Patients in this group will only undergo sural nerve and muscle biopsy
  Interventions: Procedure: Biopsy Alone
- Biopsy and RPNI (Experimental): Patients in this group will undergo RPNI during their sural nerve and muscle biopsy
  Interventions: Procedure: Peripheral Nerve Regenerative Interface (RPNI) and Nerve/Muscle Biopsy

INTERVENTIONS:
Procedure: Peripheral Nerve Regenerative Interface (RPNI) and Nerve/Muscle Biopsy — RPNI is a surgical technique which wraps denervated muscle targets around severed nerve ends.
  Arms: Biopsy and RPNI
Procedure: Biopsy Alone — Sural nerve and muscle biopsy performed in the standard fashion.
  Arms: Biopsy Alone

SUMMARY:
The purpose of our project is to determine if incorporating preventative surgical techniques such as regenerative peripheral nerve interfaces (RPNI) into sural nerve biopsy can reduce the incidence of symptomatic neuroma formation. Findings from this study will inform best practice guidelines and can dramatically impact patient care, improve patient quality of life, and reduce the number of required repeat operations.

DETAILED DESCRIPTION:
Neuromas are a known complication from traumatic injury or surgery, including nerve biopsies. Neuromas are formed by non-neoplastic aberrant proliferation of injured nerves that cannot innervate an end target resulting in a neuroma bulb made of free nerve ends, fibrotic tissue, and blood vessels. Neuromas can cause significant, debilitating pain resulting in decreased quality of life for patients and potential repeat operative interventions. The incidence rate of neuroma formation following injury is not well described but previous literature reports rates up to 30% with 14% of patients requiring repeat operation. In order to address this problem, numerous preventative and therapeutic measures have been explored. Nonsurgical management options such as desensitization, anesthetic and/or steroid injections, analgesia, and nerve stimulation have yielded mixed results.10 Therefore there is a need for reproducible and reliable prevention and treatment strategies for painful neuroma. Currently, the main surgical interventions consist of targeted muscle reinnervation (TMR) and regenerative peripheral nerve interface (RPNI). In TMR, free nerve ends are transferred onto recipient motor nerves, whereas in RPNI, free nerve ends are wrapped in a free muscle graft. Both methods provide denervated muscle targets for nerve ends. Compared to TMR, and other microsurgical measures such as primary repair or nerve grafting, RPNI is a much simpler operation that can easily be performed in the minor procedures or ward setting where nerve biopsies are usually completed. Given the functional impact from painful neuromas and subsequent burden on operative resources, efforts should be taken to prevent neuroma formation with RPNI at time of biopsy. Our project could directly improve patient care by substantiating the need for preventative measures for neuroma formation during for sural nerve biopsy thereby changing the standard of care. Given the significant pain, decreased quality of life, and need for repeat interventions, incorporating RPNI could have dramatic impacts on patient care and reduce operative and resources burdens.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old and older who are referred for sural nerve and muscle biopsy to the University of British Columbia Division of Plastic Surgery from January 2025 onwards for diagnostic or prognostic clarification of a medical condition.

Exclusion Criteria:

* Patients with previous nerve trauma (traumatic injury, surgery, or repeat biopsy) of biopsied nerve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Symptomatic neuroma formation (sensation) | 6 months post-op
  Change From Baseline in Subjective Sensation on a 10-Point Scale at 6 Months
Symptomatic neuroma formation (pain) | 6 months
  Change From Baseline in Pain Scores on the Numerical Pain Rating Scale at 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jenna-Lynn Senger, MD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - UBC Division of Plastic Surgery, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Saint Pauls Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lans J, Gamo L, DiGiovanni CW, Chen NC, Eberlin KR. Etiology and Treatment Outcomes for Sural Neuroma. Foot Ankle Int. 2019 May;40(5):545-552. doi: 10.1177/1071100719828375. Epub 2019 Feb 2. PMID 30712380
- [Background] Radtke C, Kocsis JD, Reimers K, Allmeling C, Vogt PM. Sural nerve defects after nerve biopsy or nerve transfer as a sensory regeneration model for peripheral nerve conduit implantation. Med Hypotheses. 2013 Sep;81(3):500-2. doi: 10.1016/j.mehy.2013.06.020. Epub 2013 Jul 16. PMID 23867139
- [Background] Ducic I, Yoon J, Buncke G. Chronic postoperative complications and donor site morbidity after sural nerve autograft harvest or biopsy. Microsurgery. 2020 Sep;40(6):710-716. doi: 10.1002/micr.30588. Epub 2020 Apr 10. PMID 32277511
- [Background] Hilton DA, Jacob J, Househam L, Tengah C. Complications following sural and peroneal nerve biopsies. J Neurol Neurosurg Psychiatry. 2007 Nov;78(11):1271-2. doi: 10.1136/jnnp.2007.116368. Epub 2007 Jun 5. PMID 17550992
- [Background] Chang BL, Mondshine J, Fleury CM, Attinger CE, Kleiber GM. Incidence and Nerve Distribution of Symptomatic Neuromas and Phantom Limb Pain after Below-Knee Amputation. Plast Reconstr Surg. 2022 Apr 1;149(4):976-985. doi: 10.1097/PRS.0000000000008953. PMID 35188944
- [Background] Aslami ZV, Leland CR, Strike SA, Forsberg JA, Morris CD, Levin AS, Tuffaha SH. Symptomatic Neuroma Development following En Bloc Resection of Skeletal and Soft-Tissue Tumors: A Retrospective Analysis of 331 Cases. Plast Reconstr Surg. 2024 Apr 1;153(4):873-883. doi: 10.1097/PRS.0000000000010659. Epub 2023 May 18. PMID 37199679
- [Background] Cychosz CC, Eisenberg J, Glass N, Fleury I, Buckwalter V JA, Phisitkul P, Femino JE. Outcomes of Surgical Treatment for Sural Neuritis: A Retrospective Case Series. Foot Ankle Int. 2023 Sep;44(9):845-853. doi: 10.1177/10711007231184472. Epub 2023 Jul 21. PMID 37477149
- [Background] Leach GA, Dean RA, Kumar NG, Tsai C, Chiarappa FE, Cederna PS, Kung TA, Reid CM. Regenerative Peripheral Nerve Interface Surgery: Anatomic and Technical Guide. Plast Reconstr Surg Glob Open. 2023 Jul 17;11(7):e5127. doi: 10.1097/GOX.0000000000005127. eCollection 2023 Jul. PMID 37465283
- [Background] Yang H, Dong Y, Wang Z, Lai J, Yao C, Zhou H, Alhaskawi A, Hasan Abdullah Ezzi S, Kota VG, Hasan Abdulla Hasan Abdulla M, Lu H. Traumatic neuromas of peripheral nerves: Diagnosis, management and future perspectives. Front Neurol. 2023 Jan 11;13:1039529. doi: 10.3389/fneur.2022.1039529. eCollection 2022. PMID 36712443
- [Background] Hooper RC, Cederna PS, Brown DL, Haase SC, Waljee JF, Egeland BM, Kelley BP, Kung TA. Regenerative Peripheral Nerve Interfaces for the Management of Symptomatic Hand and Digital Neuromas. Plast Reconstr Surg Glob Open. 2020 Jun 4;8(6):e2792. doi: 10.1097/GOX.0000000000002792. eCollection 2020 Jun. PMID 32766027
- [Background] Vlot MA, Wilkens SC, Chen NC, Eberlin KR. Symptomatic Neuroma Following Initial Amputation for Traumatic Digital Amputation. J Hand Surg Am. 2018 Jan;43(1):86.e1-86.e8. doi: 10.1016/j.jhsa.2017.08.021. Epub 2017 Sep 23. PMID 28951100
- [Background] Wang Z, Yi XZ, Yu AX. Regenerative peripheral nerve interface prevents neuroma formation after peripheral nerve transection. Neural Regen Res. 2023 Apr;18(4):814-818. doi: 10.4103/1673-5374.353498. PMID 36204848
- [Background] van der Avoort DJ, Hovius SE, Selles RW, van Neck JW, Coert JH. The incidence of symptomatic neuroma in amputation and neurorrhaphy patients. J Plast Reconstr Aesthet Surg. 2013 Oct;66(10):1330-4. doi: 10.1016/j.bjps.2013.06.019. Epub 2013 Jul 8. PMID 23845907
- [Background] Wolvetang NHA, Lans J, Verhiel SHWL, Notermans BJW, Chen NC, Eberlin KR. Surgery for Symptomatic Neuroma: Anatomic Distribution and Predictors of Secondary Surgery. Plast Reconstr Surg. 2019 Jun;143(6):1762-1771. doi: 10.1097/PRS.0000000000005664. PMID 30907815
- [Background] Senger JL, Thorkelsson A, Wang BY, Chan KM, Kemp SWP, Webber CA. Comparison of 2 Regenerative Peripheral Nerve Interface Techniques for the Treatment of Rat Neuroma Pain. Plast Reconstr Surg. 2024 Aug 1;154(2):346-349. doi: 10.1097/PRS.0000000000010911. Epub 2023 Jul 4. PMID 37400949
- [Background] Mauch JT, Kao DS, Friedly JL, Liu Y. Targeted muscle reinnervation and regenerative peripheral nerve interfaces for pain prophylaxis and treatment: A systematic review. PM R. 2023 Nov;15(11):1457-1465. doi: 10.1002/pmrj.12972. Epub 2023 May 28. PMID 36965013
- [Background] Santosa KB, Oliver JD, Cederna PS, Kung TA. Regenerative Peripheral Nerve Interfaces for Prevention and Management of Neuromas. Clin Plast Surg. 2020 Apr;47(2):311-321. doi: 10.1016/j.cps.2020.01.004. Epub 2020 Feb 1. PMID 32115057
- [Background] Hu Y, Ursu DC, Sohasky RA, Sando IC, Ambani SLW, French ZP, Mays EA, Nedic A, Moon JD, Kung TA, Cederna PS, Kemp SWP, Urbanchek MG. Regenerative peripheral nerve interface free muscle graft mass and function. Muscle Nerve. 2021 Mar;63(3):421-429. doi: 10.1002/mus.27138. Epub 2020 Dec 20. PMID 33290586
- [Background] Schoeller T, Huemer GM, Shafighi M, Gurunluoglu R, Wechselberger G, Piza-Katzer H. Microsurgical repair of the sural nerve after nerve biopsy to avoid associated sensory morbidity: a preliminary report. Neurosurgery. 2004 Apr;54(4):897-900; discussion 900-1. doi: 10.1227/01.neu.0000114143.07529.a6. PMID 15046656
- [Background] Kang J, Yang P, Zang Q, He X. Traumatic neuroma of the superficial peroneal nerve in a patient: a case report and review of the literature. World J Surg Oncol. 2016 Sep 10;14(1):242. doi: 10.1186/s12957-016-0990-6. PMID 27613606